CLINICAL TRIAL: NCT06051305
Title: Flexible Attention Sensory Training for Youth with Chronic Pain: a Feasibility and Acceptability Study
Brief Title: Flexible Attention Sensory Training for Youth with Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Laura E Simons, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 67616
Record Dates: First submitted 2023-08-16; First posted 2023-09-22 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Persistent Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sensory Training (Experimental): Daily protocol - gamified sensory training
  Interventions: Behavioral: Sensory Training

INTERVENTIONS:
Behavioral: Sensory Training — Participants will use gamified sensory training technology once daily for 8 weeks. This will involve participants completing a 15 minute sensory training session using the provided technology. The tool used in this study has two components. The first is a game that can be downloaded onto any smartphone device. The second component is two tactile devices that can be attached to the body.

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of gamified sensory rehabilitation training technology for children with chronic musculoskeletal pain.

DETAILED DESCRIPTION:
The TrainPain devices allows patients with chronic pain to perform sensory rehabilitation training at home, in a gamified format. The system uses a temporary tactile discrimination task, which directly engages inhibitory functions of the somatosensory cortex. In this way, the game trains the brain's sensory system to be more precise. The technology's dual-probe system allows sensory stimuli to be delivered to multiple body locations, which trains patients to flexibly shift their attention towards and away from pain according to dynamic game-directed goals. The sensory training reduces hypervigilance towards painful body regions and enables flexible attention shifting to engage with daily goals. Last, the TrainPain system captures and quantifies performance over time, providing a breadth of intricate and precise data, thus allowing the research team to assess outcomes and mechanisms of training effects. In preliminary studies with adults, TrainPain is shown to be highly engaging, and effective at reducing pain in adults with widespread musculoskeletal (MSK) pain. The current pilot study intends to establish, for the first time, the feasibility and acceptability of using the TrainPain system among youth with chronic MSK pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of musculoskeletal pain including chronic regional pain syndrome
* English speaking

Exclusion Criteria:

* Diagnosis of neurological conditions such as seizures, cerebral palsy, developmental delay
* Severe affect disorders (e.g. severe depression/anxiety) from medical record review
* Chronic skin disease or topical allergies that would be worsened by the use of sensor tape

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Acceptability of the Intervention- Net Promoter Score | Discharge (at 8 weeks)
  Acceptability will be evaluated by examining mean promoter score (measured on 10-point Likert scale) post intervention. Range 0-10 (higher scores indicate more acceptability). Questionnaire will be administered to youth with chronic pain.
Acceptability of the Intervention- Qualitative Interview | Discharge (at 8 weeks)
  Acceptability will also be assessed qualitatively at the end of treatment through interview questions related to acceptability, ease of use, comprehensibility, and suggestions for improvement. Survey responses will be reported categorically. Qualitative responses will be described and summarized.
Acceptability of the Intervention- Theoretical framework of acceptability (TFA) Questionnaire | Discharge (at 8 weeks)
  Acceptability will also be assessed quantitatively at the end of treatment through a brief survey related to acceptability, ease of use, comprehensibility, and suggestions for improvement. Survey responses will be reported categorically. Responses are measured using a five-point Likert scale from 'Strongly disagree' to 'Strongly agree' with higher scores indicating greater acceptability.
Feasibility of the Intervention- Usage Metrics | Baseline through discharge (at 8 weeks)
  Engagement will be assessed via collected use metrics (e.g. how long the app was played each day).

SECONDARY OUTCOMES:
Brief Pain Inventory Short Form (BPI) | Baseline through discharge (at 8 weeks) weekly and follow up (1-month)
  The Brief Pain Inventory evaluates the severity of a patient's pain and the impact of this pain on the patient's daily functioning. Measured on a 10-point Likert scale (range 0-10), higher scores indicate greater pain interference. Questionnaire will be administered to youth with chronic pain.
Bodily Threat Monitoring Scale (BTMS) | Baseline, discharge (at 8 weeks), and follow up (1-month)
  Bodily threat monitoring will be assessed via a 19-item self-report measure. Higher scores indicate greater propensity to monitor the body for threatening signs and symptoms.
Patient Global Impression of Change (PGIC) Scale | Baseline, discharge (at 8 weeks), and follow up (1-month)
  Single question asking participants to rate how their condition has changed since a specified point in time, with lower scores indicating greater degree of improvement.
Pain Vigilance and Awareness Questionnaire (PVAQ) | Baseline, discharge (at 8 weeks), and follow up (1-month)
  The PVAQ is a 16-item measure of attention to pain. Participants are asked to consider behavior over the past 2-weeks and indicate how frequently (0, never; 5, always) an item was true. Higher scores indicate higher pain vigilance and awareness.
Child Pain Acceptance Questionnaire (CPAQ) | Baseline, discharge (at 8 weeks), and follow up (1-month)
  Child report on the Chronic Pain Acceptance Questionnaire for Adolescents-short form will be used to assess pain acceptance in the child. The CPAQ is an 8-item measure consisting of two subscales: Activity Engagement (4 items) and Pain Willingness (4 items). Items are rated on a 5-point Likert scale ranging from 0 (Never True) to 4 (Always True) and yield a total score for each subscale ranging from 0-16. Higher scores indicate greater Activity Engagement and greater Pain Willingness.
Multidimensional Assessment of Interoceptive Awareness Youth (MAIA-Y) | Baseline, discharge (at 8 weeks), and follow up (1-month)
  The MAIA-Y is an 8-scale state-trait questionnaire with 32 items. It measures multiple dimensions of interoception. Scoring is at the individual scale-level, with higher scores equated with more bodily sensation awareness. The individual score is also given as a percentile relative to normative sample, with extreme percentiles (>10, 90<) of clinical significance. Three scales from this measures are being administered: Attention Regulation, Self-Regulation, Trusting.
Revised Life Orientation Test (LOT-R) | Baseline, discharge (at 8 weeks), and follow up (1-month)
  The Revised Life Orientation Test will be used to assess self-reported optimism in the child. The LOT-R is a 10-item measure yielding a total score ranging from 0-20 (only 5 items are utilized in the final score calculation). Higher scores indicate greater optimism.
Childrens Hope Scale (CHS) | Baseline, discharge (at 8 weeks), and follow up (1-month)
  The Childrens Hope Scale will be used to assess self-reported hope in the child. The CHS is a 6-item measure yielding a total score ranging from 0-36, with higher scores indicating greater hope/
Pain Catastrophizing Scale (PCS-C) | Baseline, discharge (at 8 weeks), and follow up (1-month)
  The Pain Catastrophizing Scale -Child Version (PCS-C, Crombez et al., 2003) assesses negative cognitions associated with pain. The PCS-C is comprised of 13-items rated on a 5-point Likert scale (0= "not at all true" to 4 "very true"). A total score (0-52) is obtained by summing all items. Higher scores indicate higher levels of catastrophic thinking.
Weekly Diary | Treatment (weekly for 8 weeks)
  We are administering an additional 13-item weekly diary, developed by our group, which measure self-reported fear, avoidance, functioning, activity engagement, pain reactivity, and attention.
Parent Psychological Flexibility Questionnaire (PPF-P) | Baseline, discharge (at 8 weeks), and follow up (1-month)
  The Parent Psychological Flexibility Questionnaire (PPFQ-10, Timmers et al., 2019) is a 10-item parent self-report questionnaire assessing a parent's ability to accept their own distress and respond adaptively and flexibly to their child's pain. Items are rated on a 5-point Likert scale (0= " never true" to 4 = "always true") and are summed to create a total score, ranging from 0 - 40. Higher scores indicate greater parent psychological flexibility.
Pain Catastrophizing Scale (PCS-P) | Baseline, discharge (at 8 weeks), and follow up (1-month)
  Pain Catastrophizing Scale-Parent Version (PCS-P, Goubert et al., 2006) assesses parents' negative cognitions associated with their child's pain. It is comprised of 13 items rated on a 5-point Likert scale (0 = "not true at all" to 4 = "very true"). A total score (0-52) is derived by summing items, with higher scores indicating higher levels of catastrophic thinking.

OTHER OUTCOMES:
Adverse events | Baseline through 8 weeks
Treatment Expectancy and Credibility (TEC) | Baseline, discharge (at 8 weeks)
  Participants (child) and parent expectations for treatment will be measured by the Treatment Expectancy and Creditability. The TEC is comprised of 6 items rated on a 0 to 10 Likert-scale assessing expectations related to the effectiveness of the current treatment. The TEC is completed by the patient at the end of the first treatment session and at the end of treatment (8 weeks). Higher scores indicate greater expectations for treatment effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Simons, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Pediatric Pain Clinic, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borkovec, T. D., & Nau, S. D. (1972). Credibility of analogue therapy rationales. Journal of behavior therapy and experimental psychiatry, 3(4), 257-260.
- [Background] Sekhon M, Cartwright M, Francis JJ. Development of a theory-informed questionnaire to assess the acceptability of healthcare interventions. BMC Health Serv Res. 2022 Mar 1;22(1):279. doi: 10.1186/s12913-022-07577-3. PMID 35232455
- [Background] Mendoza T, Mayne T, Rublee D, Cleeland C. Reliability and validity of a modified Brief Pain Inventory short form in patients with osteoarthritis. Eur J Pain. 2006 May;10(4):353-61. doi: 10.1016/j.ejpain.2005.06.002. Epub 2005 Jul 26. PMID 16051509
- [Background] Mesaroli G, Campbell F, Hundert A, Birnie KA, Sun N, Davidge KM, Lalloo C, Davies-Chalmers C, Harris L, Stinson J. Development of a Screening Tool for Pediatric Neuropathic Pain and Complex Regional Pain Syndrome: Pediatric PainSCAN. Clin J Pain. 2021 Oct 12;38(1):15-22. doi: 10.1097/AJP.0000000000000993. PMID 34636750
- [Background] Ferguson, L., & Scheman, J. (2009). Patient global impression of change scores within the context of a chronic pain rehabilitation program. The Journal of Pain, 10(4), S73.
- [Background] Roelofs J, Peters ML, McCracken L, Vlaeyen JWS. The pain vigilance and awareness questionnaire (PVAQ): further psychometric evaluation in fibromyalgia and other chronic pain syndromes. Pain. 2003 Feb;101(3):299-306. doi: 10.1016/S0304-3959(02)00338-X. PMID 12583873
- [Background] Vowles KE, McCracken LM, McLeod C, Eccleston C. The Chronic Pain Acceptance Questionnaire: confirmatory factor analysis and identification of patient subgroups. Pain. 2008 Nov 30;140(2):284-291. doi: 10.1016/j.pain.2008.08.012. Epub 2008 Sep 27. PMID 18824301
- [Background] Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A. The Multidimensional Assessment of Interoceptive Awareness (MAIA). PLoS One. 2012;7(11):e48230. doi: 10.1371/journal.pone.0048230. Epub 2012 Nov 1. PMID 23133619
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Castarlenas E, Jensen MP, von Baeyer CL, Miro J. Psychometric Properties of the Numerical Rating Scale to Assess Self-Reported Pain Intensity in Children and Adolescents: A Systematic Review. Clin J Pain. 2017 Apr;33(4):376-383. doi: 10.1097/AJP.0000000000000406. PMID 27518484
- [Background] Gauntlett-Gilbert J, Alamire B, Duggan GB. Pain Acceptance in Adolescents: Development of a Short Form of the CPAQ-A. J Pediatr Psychol. 2019 May 1;44(4):453-462. doi: 10.1093/jpepsy/jsy090. PMID 30496433